CLINICAL TRIAL: NCT00675402
Title: Micro- and Macrovascular Adaptations in Patients With Peripheral Arterial Disease During Supervised Exercise Therapy: a MRI Study
Brief Title: Micro- and Macrovascular Adaptations in Patients With Peripheral Arterial Disease During Supervised Exercise Therapy
Acronym: VAPAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Bas Versluis, Maastricht University Hospital, dep. of Radiology
Other Study IDs: MEC 08-2-032
Record Dates: First submitted 2008-05-06; First posted 2008-05-09 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: PAOD (Peripheral Arterial Obstructive Disease)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients referred to the vascularsurgeon with complaints of claudication for their first time, will be asked to participate with the study, with respect toward the in- and exclusion criteria.
  Interventions: Other: supervised treadmill exercise program

INTERVENTIONS:
Other: supervised treadmill exercise program — Supervised treadmill therapy consists of a walking exercise on a treadmill under supervision of a physiotherapist, 2-3 times a week. This program is combined with individual walking every other day and the total duration of the program is 6 months. Guided by the painfree walking distance, every month the angle and/or speed of the treadmill will increase. A standardized protocol for this type of therapy is already in use by many physiotherapists in Limburg (Willigendael, 2005).

SUMMARY:
Given that previous studies demonstrated the feasibility of the required MRI techniques, we propose to study the macro- and microvascular adaptations in PAOD patients undergoing supervised exercise therapy. It is expected to provide valuable insights into the contribution of each vascular mechanism to the rehabilitation and to identify which vascular mechanism fails or is insufficient for a successful rehabilitation. Improvement of future treatment requires the identification of relevant adaptive mechanisms. With this we will provide early noninvasive MRI readout tools to diagnose and monitor the potential rehabilitation during any form of therapy for PAOD that affects the peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication according to a positive Rose-Edingburgh questionnaire
* Rest ankle-brachial pressure index (ABPI) < 0,90 or 10% decline in ABPI after exercise
* Arterial stenosis/occlusion of femoro-popliteal territory according to duplex/MRA measurements
* Able to ondergo exercise therapy

Exclusion Criteria:

* Chronic or acute critical ischemia
* Treated by or planned for vascular surgery or percutaneous transluminal angioplasty
* Recent onset <2 months
* Unable to perform treadmill exercise
* Diabetes mellitus
* Contra-indications for (Gadolinium-enhanced) MRI or thigh cuff inflation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the vascular surgeon with complaints of claudication for their first time, will be asked to participate with the study, with respect toward the in- and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: WH Backes, PhD, Principal Investigator — Maastricht University Hospital, dep. of Radiology
Locations (1):
- Maastricht University Hospital, Maastricht, Limburg, Netherlands